CLINICAL TRIAL: NCT03035773
Title: Simplifying Survivorship Care Planning; Comparing the Efficacy and Patient-Centeredness of Three Care Delivery Models
Brief Title: Simplifying Survivorship Care Planning
Acronym: SSCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: J16117; IRB00110605 (Other: JHMIRB); R-1410-24904 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institution)
Record Dates: First submitted 2016-12-13; First posted 2017-01-30 (Estimated); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: Oncology; Survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM A; Care Plan Only (Experimental): SCP document delivered to the patient & Primary Care Provider
  Interventions: Behavioral: Care Plan Only
- ARM B; Care Plan During Visit (Experimental): SCP document provided to the patient in an in-person survivorship visit and copy sent to PCP
  Interventions: Behavioral: Care Plan During a Visit
- ARM C; Care Plan During Visit + Additional Visit (Experimental): SCP document provided to the patient in an in-person survivorship visit with an additional follow-up visit and copy of the document sent to PCP
  Interventions: Behavioral: Care Plan During a Visit with an Additional Visit

INTERVENTIONS:
Behavioral: Care Plan Only — Patient participants randomized to Arm A will be sent a copy of the SCP within 3 months of completion of treatment and a copy will be added to their medical record. A copy of the SCP will also be sent to the PCP on record. The SCP will be completed by a nurse, nurse practitioner, or physician assistant. The SCP will be accompanied by a cover letter that will be signed by a member of the clinical team.
  Other Names: Arm A
  Arms: ARM A; Care Plan Only
Behavioral: Care Plan During a Visit — Patient participants randomized to Arm B will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider on record. The visit will be scheduled after consent is signed and will occur between 1 and 3 months after completion of treatment. The visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues.
  Other Names: Arm B
  Arms: ARM B; Care Plan During Visit
Behavioral: Care Plan During a Visit with an Additional Visit — Participants randomized to Arm C will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider. The visit will be scheduled after consent is signed and will occur between 1-3 months after completion of treatment. The initial visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues. Patients will also receive a follow up survivorship visit 7-10 months after the end of treatment that will focus on a review of the SCP and offer the opportunity to ask about any persistent or emerging issues.
  Other Names: Arm C
  Arms: ARM C; Care Plan During Visit + Additional Visit

SUMMARY:
OBJECTIVE: The purpose of this study is to identify an SCP process that is patient-centered, effective in promoting appropriate survivorship care and can be successfully implemented for patients with different types of cancer who are being treated in a broad range of clinical settings. There is a need for research related to SCP that prioritizes outcomes that are most highly valued by patients, caregivers and clinical stakeholders.

DETAILED DESCRIPTION:
BACKGROUND: Each year, approximately 1.6 million people are diagnosed with cancer and the relative 5-year survival rate across all cancer types approaches 70%. As of 2014, there were almost 15 million Americans living with a history of cancer. Cancer survivors face a variety of health care needs, including surveillance for recurrence, treatment for long-term and late effects of cancer and its treatment, general primary and preventive care, management of any comorbidities, encouragement of healthy lifestyle behaviors, and attention to psychosocial issues. In 2005, the Institute of Medicine (IOM) report 'From Cancer Patient to Cancer Survivor: Lost in Transition' highlighted the challenges that cancer survivors face as they transition from acute treatment. The completion of acute cancer treatment is a critical juncture at which patients are in need of better support and communication to ensure optimal health and quality of life outcomes as they transition to long-term survivorship. Cancer survivors face substantial deficiencies in the quality of care that they receive, including both underuse of recommended care and overuse of services that are not recommended for routine follow-up. The 2005 IOM report called for all patients completing acute treatment to be provided with a survivorship care plan (SCP) that summarizes treatments received and outlines future healthcare priorities in order to facilitate effective management of health care between survivors and their oncology and primary care providers.

STUDY PROCEDURES: The primary aim of this trial is to assess whether there is a difference among three SCP models of varying levels of resource intensity and patients' receipt of recommended health services in the months following completion of acute treatment. The investigators will conduct a randomized controlled trial (RCT) to measure whether the provision of the SCP to the survivor and primary care provider (PCP) is associated with survivors' receipt of cancer follow-up care as outlined on their SCP (primary outcome). Avoidance of non-recommended care, receipt of recommended primary and preventive care, and patient-reported outcome measures will serve as secondary endpoints.

Participants in the RCT will have been treated for breast, prostate, or colorectal cancer. This RCT will be conducted in four oncology clinics in two medical systems. The investigators will enroll survivors of Stage I-III breast, prostate, or colorectal cancer who are completing treatment and transitioning to long-term survivorship, and use a stratified randomization to assign participants to one of three study conditions (Arms A, B or C). This study will focus specifically on the period following completion of acute treatment (e.g., surgery, radiation, and chemotherapy); patients receiving long-term adjuvant endocrine/antibody therapies will also be eligible.

The proposed trial will be conducted at Johns Hopkins Medical Institution (JHMI) and Peninsula Regional Medical Center (PRMC). JHMI is a large, academic medical center in an urban setting with distinct treatment programs based on disease site. At JHMI, the investigators will recruit from the Breast Cancer Program, the Genitourinary Cancer Program (prostate cancer), and Gastrointestinal Cancer Program (colorectal cancer). These programs operate across disciplines (e.g., medical, radiation, and surgical oncology) but separately from each other, enabling evaluation of 3 separate clinical settings within JHMI. In addition, the trial will include the PRMC Richard A. Henson Cancer Institute, a community cancer program located in the rural area of Maryland's eastern shore. At PRMC there is a single general oncology practice. The four programs differ in the extent to which survivorship care planning is already a part of routine care. As yet, none of the clinics in this study has a consistent format for the delivery of SCP universally at the completion of acute treatment. The study design (cancer types, clinical systems and SCP models) is intended to enable the development of real-world best practices for the implementation of SCPs and assess whether these are consistent or vary across a wide range of clinical contexts and survivor characteristics.

Each participant will be followed for 18 months, with the number of visits dependent on the randomization arm (described below). The investigators will abstract 18 months of follow-up data for enrolled patients from medical records, as well as from patient reports of health service use; data will be collected at months 6, 12, and 18. The investigators will obtain and abstract medical records guided by the information in the summary document (see Health Services Use Summary included as a supplemental study document) and from the patient using provided tracking tools of providers they have seen, tests they have undergone, etc. (see Tip Sheet in supplemental study documents). Patient-reported outcomes will be collected at baseline, 6, 12, and 18 months primarily via a REDCap form, with telephone or in-person data collection as a back-up when needed.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older;
* Diagnosed with breast, colorectal, or prostate cancer (stages I-III);
* Treated with intent to cure
* People who are on long-term (>1 year) chronic treatment are eligible;
* No evidence of disease;
* Able to complete the study data collection in English;
* Had their cancer care primarily managed by either JHMI or PRMC, with JHMI or PRMC primarily responsible for the patients' survivorship care; and
* Has private insurance, or covered by Medicare or Medicaid.

Exclusion Criteria:

* Younger than 21 years of age;
* Diagnosed with in situ or metastatic breast, prostate or colorectal cancer (i.e. Stage 0 or IV);
* Not treated with intent to cure;
* Did not have cancer care primarily managed within one of the 4 participating clinics, or JHMI or PRMC is not primarily responsible for the patients' survivorship care; and
* Does not have health insurance at screening.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2015-10; Primary Completion 2020-12 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Smith, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beckjord EB, Arora NK, McLaughlin W, Oakley-Girvan I, Hamilton AS, Hesse BW. Health-related information needs in a large and diverse sample of adult cancer survivors: implications for cancer care. J Cancer Surviv. 2008 Sep;2(3):179-89. doi: 10.1007/s11764-008-0055-0. Epub 2008 Jun 3. PMID 18792791
- [Background] Dunn, R., Crowley, S., & Janz, N. (2011). Impact of a transition visit on addressing quality of life and readiness to assume greater self-management among breast cancer survivors. Psycho-Oncology, 20(S1), S91.
- [Background] Gotay CC, Pagano IS. Assessment of Survivor Concerns (ASC): a newly proposed brief questionnaire. Health Qual Life Outcomes. 2007 Mar 13;5:15. doi: 10.1186/1477-7525-5-15. PMID 17352831
- [Background] Hershman DL, Greenlee H, Awad D, Kalinsky K, Maurer M, Kranwinkel G, Brafman L, Jayasena R, Tsai WY, Neugut AI, Crew KD. Randomized controlled trial of a clinic-based survivorship intervention following adjuvant therapy in breast cancer survivors. Breast Cancer Res Treat. 2013 Apr;138(3):795-806. doi: 10.1007/s10549-013-2486-1. Epub 2013 Mar 31. PMID 23542954
- [Background] Hewitt, M., Greenfield, S., & Stovall, E. (Eds.). (2005). From cancer patient to cancer survivor: lost in transition. National Academies Press.
- [Background] Kent EE, Arora NK, Rowland JH, Bellizzi KM, Forsythe LP, Hamilton AS, Oakley-Girvan I, Beckjord EB, Aziz NM. Health information needs and health-related quality of life in a diverse population of long-term cancer survivors. Patient Educ Couns. 2012 Nov;89(2):345-52. doi: 10.1016/j.pec.2012.08.014. Epub 2012 Sep 28. PMID 23021856
- [Background] Mallinger JB, Griggs JJ, Shields CG. Patient-centered care and breast cancer survivors' satisfaction with information. Patient Educ Couns. 2005 Jun;57(3):342-9. doi: 10.1016/j.pec.2004.09.009. PMID 15893218
- [Background] Nelson DE, Kreps GL, Hesse BW, Croyle RT, Willis G, Arora NK, Rimer BK, Viswanath KV, Weinstein N, Alden S. The Health Information National Trends Survey (HINTS): development, design, and dissemination. J Health Commun. 2004 Sep-Oct;9(5):443-60; discussion 81-4. doi: 10.1080/10810730490504233. PMID 15513791
- [Background] Smith KC, Tolbert E, Hannum SM, Radhakrishnan A, Zorn K, Blackford A, Greco S, Smith K, Snyder CF. Comparing Web-Based Provider-Initiated and Patient-Initiated Survivorship Care Planning for Cancer Patients: A Randomized Controlled Trial. JMIR Cancer. 2016 Aug 30;2(2):e12. doi: 10.2196/cancer.5947. PMID 28410187

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM A (Care Plan Only): SCP document delivered to the patient & Primary Care Provider
  Care Plan Only: Patient participants randomized to Arm A will be sent a copy of the SCP within 3 months of completion of treatment and a copy will be added to their medical record. A copy of the SCP will also be sent to the PCP on record. The SCP will be completed by a nurse, nurse practitioner, or physician assistant. The SCP will be accompanied by a cover letter that will be signed by a member of the clinical team.
- ARM B (Care Plan During a Visit): SCP document provided to the patient in an in-person survivorship visit and copy sent to PCP
  Care Plan During a Visit: Patient participants randomized to Arm B will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider on record. The visit will be scheduled after consent is signed and will occur between 1 and 3 months after completion of treatment. The visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues.
- ARM C (Care Plan During a Visit With an Additional Visit): SCP document provided to the patient in an in-person survivorship visit with an additional follow-up visit and copy of the document sent to PCP
  Care Plan During a Visit with an Additional Visit: Participants randomized to Arm C will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider. The visit will be scheduled after consent is signed and will occur between 1-3 months after completion of treatment. The initial visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues. Patients will also receive a follow up survivorship visit 7-10 months after the end of treatment that will focus on a review of the SCP and offer the opportunity to ask about any persistent or emerging issues.
Period: Overall Study
Arm/Group | ARM A (Care Plan Only) | ARM B (Care Plan During a Visit) | ARM C (Care Plan During a Visit With an Additional Visit)
Started | 126 | 125 | 127
Completed | 107 | 105 | 104
Not Completed | 19 | 20 | 23

BASELINE CHARACTERISTICS:
Groups:
- ARM A - Care Plan Only: SCP document delivered to the patient & Primary Care Provider
  Care Plan Only: Patient participants randomized to Arm A will be sent a copy of the SCP within 3 months of completion of treatment and a copy will be added to their medical record. A copy of the SCP will also be sent to the PCP on record. The SCP will be completed by a nurse, nurse practitioner, or physician assistant. The SCP will be accompanied by a cover letter that will be signed by a member of the clinical team.
- ARM B - Care Plan During a Visit: SCP document provided to the patient in an in-person survivorship visit and copy sent to PCP
  Care Plan During a Visit: Patient participants randomized to Arm B will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider on record. The visit will be scheduled after consent is signed and will occur between 1 and 3 months after completion of treatment. The visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues.
- ARM C - Care Plan During a Visit With an Additional Visit: SCP document provided to the patient in an in-person survivorship visit with an additional follow-up visit and copy of the document sent to PCP
  Care Plan During a Visit with an Additional Visit: Participants randomized to Arm C will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider. The visit will be scheduled after consent is signed and will occur between 1-3 months after completion of treatment. The initial visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues. Patients will also receive a follow up survivorship visit 7-10 months after the end of treatment that will focus on a review of the SCP and offer the opportunity to ask about any persistent or emerging issues.
- Total: Total of all reporting groups
Arm/Group | ARM A - Care Plan Only | ARM B - Care Plan During a Visit | ARM C - Care Plan During a Visit With an Additional Visit | Total
Number analyzed (Participants) | 126 | 125 | 127 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.6) | 61.5 (12.0) | 60.8 (12.1) | 61.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 66 | 64 | 192
  Male | 64 | 59 | 63 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 4 | 13
  Not Hispanic or Latino | 120 | 122 | 123 | 365
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 28 | 23 | 75
  White | 97 | 97 | 98 | 292
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 126 | 125 | 127 | 378

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Compliant With Follow-up Care Visits
Description: The primary outcome classifies patients as compliant or non-compliant based on whether they were compliant on all visits, tests/procedures, and non-oral medication recommendations included in their care plans.
Time Frame: 18 Months
Population: The primary analysis was by intention to treat. To be included, participants had to have received an SCP and have data from 18 months of follow-up.
  Four patients (3 from Arm A and 1 from ARM C) were not included in the primary outcome analysis because there were no recommendations listed in their care plans.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM A - Care Plan Only | ARM B - Care Plan During a Visit | ARM C - Care Plan During a Visit With an Additional Visit
Number analyzed (Participants) | 104 | 105 | 103
Participants | 47 | 53 | 44

2. Secondary Outcome: Number of Participants Who Received an Annual Physical Exam
Description: This secondary outcome classifies participants as having had an annual physical exam based on medical record review. This outcome was operationalized as a dichotomous variable (received recommended primary care: yes/no). Participants were included in this analysis if they had a primary care visit recommended on their survivorship care plan.
Time Frame: 18 Months
Measure: Count of Participants; unit: Participants
Arm/Group | ARM A; Care Plan Only | ARM B; Care Plan During Visit | ARM C; Care Plan During Visit + Additional Visit
Number analyzed (Participants) | 66 | 56 | 61
Participants | 48 | 40 | 43

3. Secondary Outcome: Number of Participants Who Received Tests and Procedures Recommended on Their Survivorship Care Plan
Description: These data are generated through electronic medical record review. This outcome is operationalized as a dichotomous variable (received recommended tests and procedures: yes/no).
Time Frame: 18 Months
Population: Only participants who had any tests or procedures recommended on their personalized survivorship care plan were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | ARM A; Care Plan Only | ARM B; Care Plan During Visit | ARM C; Care Plan During Visit + Additional Visit
Number analyzed (Participants) | 104 | 101 | 100
Participants | 82 | 78 | 73

4. Secondary Outcome: Number of Participants Who Received Cancer-related Tests Consistent With Overuse
Description: This analysis compared potential overuse of surveillance tests between cancer types (breast, prostate and colorectal). This outcome will be operationalized as a dichotomous variable (did not receive inappropriate care: yes/no). The outcome relates to participants who received care not specified on their care plan and on a guideline predetermined list of "not recommended surveillance. This was determined through a physician chart review.
Time Frame: 18 Months
Population: Only participants with a history of breast, colorectal, or prostate cancer were analyzed. The protocol specified that this analysis would be by cancer type, not study arm as surveillance tests analyzed were not specified on survivorship care plans.
Measure: Count of Participants; unit: Participants
Groups:
- Breast Cancer: Participants with a history of breast cancer
- Colorectal Cancer: Participants with a history of colorectal cancer
- Prostate Cancer: Participants with a history of prostate cancer
Arm/Group | Breast Cancer | Colorectal Cancer | Prostate Cancer
Number analyzed (Participants) | 137 | 67 | 112
Participants | 22 | 0 | 1

5. Secondary Outcome: Patient-reported Outcomes: Preparing for Life as a (New) Survivor (PLANS)
Description: PLANS is a cancer survivorship questionnaire with 2 items specifically related to survivorship care planning. These items are 'I feel prepared for what to expect over the next year' (score range 1-4 with 4 being a more positive score) and 'There is a well-coordinated plan for my cancer care' (score range 1-10 with 1 being "Not at all confident and 10 being "Extremely confident".
Time Frame: 18 Months
Population: Analysis includes participants who completed the PLANS data at 18 months post baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM A; Care Plan Only | ARM B; Care Plan During Visit | ARM C; Care Plan During Visit + Additional Visit
Number analyzed (Participants) | 71 | 71 | 69
score on a scale
  Feel prepared for what to expect in the coming year | 3.3 (0.6) | 3.2 (0.7) | 3.1 (0.7)
  There is a well-coordinated plan for your cancer care | 7.7 (1.8) | 7.4 (2.3) | 7.4 (2.3)

6. Secondary Outcome: Patient-reported Outcomes: Assessment of Survivor Concerns (ASC)
Description: The outcome is a sum score of a 5-item scale with a minimum score of 5 and a maximum score of 20 with a higher score indicating greater worry (worse outcome).
Time Frame: 18 Months
Population: Participants who completed Patient Reported Outcomes data at 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM A; Care Plan Only | ARM B; Care Plan During Visit | ARM C; Care Plan During Visit + Additional Visit
Number analyzed (Participants) | 71 | 71 | 69
score on a scale | 11.2 (3.6) | 11.2 (4.0) | 11.1 (3.5)

7. Secondary Outcome: Patient-reported Outcomes: Follow-up Care Use Among Survivors (FOCUS)-Information Needs Module
Description: Questionnaire asking about informational needs on 12 topics. Responses for each question can be yes/no/not sure. Reported the total number of health needs responded to as "yes". Outcome is a sum of reported needs. Score range from 0-12 with a higher score reflecting more informational needs.
Time Frame: 18 Months
Population: Analysis is of the participants who completed Patient Reported Outcomes data collection at 18 month timepoints
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARM A; Care Plan Only | ARM B; Care Plan During Visit | ARM C; Care Plan During Visit + Additional Visit
Number analyzed (Participants) | 71 | 71 | 69
units on a scale | 3.7 (3.4) | 3.8 (3.6) | 3.9 (3.7)

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- ARM C - Care Plan During a Visit an Additional Visit: SCP document provided to the patient in an in-person survivorship visit with an additional follow-up visit and copy of the document sent to PCP
  Care Plan During a Visit with an Additional Visit: Participants randomized to Arm C will receive a copy of the SCP during an in-person 'stethoscope free' visit with a nurse, nurse practitioner, or physician assistant. A copy of the SCP will be added to the medical record and a copy will be sent to the primary care provider. The visit will be scheduled after consent is signed and will occur between 1-3 months after completion of treatment. The initial visit will focus on review of the SCP content and offer an opportunity for patients to ask questions about any aspect of the plan or associated treatment and survivorship issues. Patients will also receive a follow up survivorship visit 7-10 months after the end of treatment that will focus on a review of the SCP and offer the opportunity to ask about any persistent or emerging issues.
Arm/Group | ARM A - Care Plan Only | ARM B - Care Plan During a Visit | ARM C - Care Plan During a Visit an Additional Visit
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/125 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/125 | 0/127
Other Adverse Events (participants affected / at risk) | 0/126 | 0/125 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03035773/Prot_SAP_000.pdf